CLINICAL TRIAL: NCT06639503
Title: Genicular Nerve Block for Analgesia After Open Reduction Internal Fixation of Tibial Plateau Fractures: A Prospective, Randomized Controlled Trial
Brief Title: Genicular Nerve Block After Open Reduction Internal Fixation of Tibial Plateau
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB23-0930
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Tibial Plateau Fractures
Keywords: peri-incisional local anesthesia; genicular nerve block; Tibial Plateau Fractures; open reduction internal fixation
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Subgroups will be determined using equal block randomization. Blocks will be set to groups of 4 with each block of 4 comprising 2 peri-incisional local anesthesia and 2 genicular nerve blockade opaque envelopes in random order.
Who Masked: Participant
Masking Description: The envelope will be opened in the operating room prior to beginning the procedure. This ensures subjects are blinded to their treatment modality.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peri-incisional local anesthesia (No Intervention): subjects randomized to peri-incisional local anesthesia administration will receive an injection of 25 ml of 0.25% bupivacaine across all incisions at the time of wound closure (standard of care)
- Genicular nerve blockade (Experimental): Subjects randomized to genicular nerve block will receive a fluoroscopic guided injection of 5 ml of 0.25% bupivacaine at the described locations of the superolateral genicular nerve, super medial genicular nerve, inferomedial genicular nerve, recurrent fibular nerve, and infrapatellar branch of the saphenous nerve under fluoroscopic guidance at the time of wound closure
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Bupivacain — 5mL 0.25% bupivacain
  Arms: Genicular nerve blockade

SUMMARY:
The investigators are conducting this research study to find better ways of treating pain following knee surgery. There is a standard (accepted) approach, which involves injection of numbing medication into the area around the participant surgical incision. The investigators hope to discover if providing numbing medication to a nerve that controls pain in a larger area of the knee (a nerve block), might be better at post-operative pain control.

DETAILED DESCRIPTION:
The investigators are conducting this research study to find better ways of treating pain following knee surgery like the one the participant will be having. There is a standard (accepted) approach, which involves injection of numbing medication into the area around the participant surgical incision. The investigators hope to discover if providing numbing medication to a nerve that controls pain in a larger area of the knee (a nerve block), might be better at post-operative pain control. This type of nerve block is commonly used to treat other knee pains, like that associated with arthritis, after knee replacements, and after repairs of the knee ligaments; however, it is considered experimental in your case, as its effects (good or bad) are unknown in the type of knee surgery the participant are undergoing.

The investigators plan is to decide at random, like the flip of a coin, whether to give numbing medication (0.25% bupivacaine) around the incision like the investigators normally would or give it instead to block the pain sensors around the knee. The participant would get medication either at the incision (shin) or the knee, depending on which arm the participant are in (research). The participant will also be given pain medication pills by your surgeon as part of the participant normal postoperative care (not research).

ELIGIBILITY:
Inclusion Criteria:

• Any adult patient (ages 18 and over) undergoing open reduction internal fixation of an acute isolated tibial plateau fracture

Exclusion Criteria:

* Subjects younger than 18
* Polytraumatized Subjects
* Subjects with pathologic fractures
* Subjects with tibial plateau fractures treated nonoperatively
* Subjects with tibial plateau fractures treated operatively but with re-operations at the same site
* Subjects with open fractures
* Subjects with fracture-dislocations
* Subjects with active or history of anxiety
* Subjects with visual analog scale anxiety score ≥ 7 measured preoperatively
* Subjects with chronic pain syndromes
* Subjects with chronic opioid use
* Subjects with illicit drug use disorder
* Subjects with alcohol abuse disorder
* Subjects with kidney disease precluding use of ketorolac
* Subjects with liver disease precluding the use of acetaminophen
* Subjects with allergy to acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), opiates or local anesthesia
* Subjects with inability to provide a visual analog scale score postoperatively
* Subjects with contraindications to receiving peripheral nerve blocks, including relevant neurologic deficits, active infection at sites of injections - re-operation at the same site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Pain Ratings from Visual Analog Scale (VAS) | one hour, two hours, and discharge from PACU
  To determine if genicular nerve blockade after open reduction internal fixation of tibial plateau fractures compared to standard care of peri-incisional local anesthetic leads to decreased pain as measured by visual analog scale at one hour postoperatively, two hours postoperatively, and at Post Anesthesia Care Unit (PACU) discharge. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')

SECONDARY OUTCOMES:
Comparing blocks | one hour after surgery, 2 hours after surgery, and discharge from PACU
  To assess the effect of genicular nerve block compared to standard peri-incisional local anesthetic on analgesic consumption in the Post Anesthesia Care Unit (PACU) using they Visual analog (VAS) scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Block effect on range of motion | PACU discharge
  To assess the effect of genicular nerve block compared to standard peri-incisional local anesthetic on postoperative function as assessed by postoperative knee range of motion at time of Post Anesthesia Care Unit (PACU) discharge.
VAS score daily first three days after surgery | daily for three days after surgery
  To determine the effect of genicular nerve block compared to standard peri-incisional local anesthetic on pain control for the first three days after surgery as measured by the visual analog scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
Brief pain inventory (short scale) daily first three days after surgery | daily first three days after surgery
  To determine the effect of genicular nerve block compared to standard peri-incisional local anesthetic on pain control for the first three days after surgery as measured by the Brief pain inventory (short scale). the brief pain inventory (Short form) uses a 0 to 10 numeric rating scales for item rating.
  1 - 4 = Mild Pain 5 - 6 = Moderate Pain 7 - 10 = Severe Pain
effect of genicular nerve blockade compared to standard peri-incisional local anesthetic | 2 weeks post surgery
  To determine the effect of genicular nerve blockade compared to standard peri-incisional local anesthetic on opiate use as determined by the number of prescription opiate pain pills remaining at 2 weeks post surgery.
Comparing blocks | daily first three days after surgery
  To assess the effect of genicular nerve block compared to standard peri-incisional local anesthetic on analgesic consumption in the Post Anesthesia Care Unit (PACU) using the Brief pain inventory (short form). the brief pain inventory (Short form) uses a 0 to 10 numeric rating scales for item rating.
  1 - 4 = Mild Pain 5 - 6 = Moderate Pain 7 - 10 = Severe Pain
Comparing blocks | 2 weeks after surgery
  To assess the effect of genicular nerve block compared to standard peri-incisional local anesthetic on analgesic consumption in the Post Anesthesia Care Unit (PACU) using opiate pill counts.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Christiano, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data